CLINICAL TRIAL: NCT06857383
Title: Assessment of Head Awareness in Chronic Migraine Patients With the Fremantle Headache Awareness Questionnaire: Turkish Version, Validity and Reliability Study
Brief Title: Head Awareness in Chronic Migraine Patients
Acronym: Awareness
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Dilara Onan, Assistant Professor, Bozok University
Other Study IDs: 2024-GOKAEK2413_2024.11.20_191
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Migraine
Keywords: migraine; awareness; headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fremantle Headache Awareness Questionnaire — It is a simple Likert-type questionnaire that evaluates individual-specific altered perception (0 = Never/Never feel like this, 1 = Rarely feel like this, 2 = Sometimes or sometimes feel like this, 3 = Often feel like this, 4 = Always or most of the time feel like this). The questionnaire asks individuals 9 questions about how they perceive their heads and headaches in relation to their bodies. The questionnaire was developed by Wand et al. in its first version as "The Fremantle Back Awareness Questionnaire". With permission from the author, the questionnaire was created by adapting the questions of the Fremantle Back Awareness Questionnaire to headache.

SUMMARY:
Research indicates that different beliefs about the nature of back problems and their future consequences direct behaviors that may cause falsely stimulated neuroplastic changes. The central nervous system can help relieve ongoing pain by regulating nociceptive activity. For this purpose, "The Fremantle Back Awareness Questionnaire" was developed to evaluate the perceptual awareness status of the back. In individuals with chronic pain, changes in body perception can be explained by the cortical reorganization that occurs in these individuals. Compared to healthy individuals, cortical thickness is reduced in the brain regions that process pain in chronic migraine patients. On the other hand, it is stated that these cortical structural changes can be reversed and recovery can be achieved by treating headache and related symptoms in chronic migraine patients. Individuals try to continue their daily lives with impaired body awareness due to pain. Decreased awareness has been studied in many neck, back and knee pain studies in the literature with Fremantle Awareness Questionnaires in different societies. In these studies, the awareness of individuals experiencing pain was found to be low and it was found that neck, waist or knee awareness was related to pain intensity, pain catastrophizing, disability, quality of life, anxiety, depression and kinesiophobia. It was even determined that awareness increased with treatments. Although reversible structural changes in the cortical regions of chronic migraine patients have been investigated with radiological imaging methods and are still being investigated, not every patient can be evaluated with radiological imaging in clinics due to cost and time problems. Therefore, a fast, practical and understandable questionnaire evaluation can benefit clinicians. When the literature is examined, there is no study evaluating the perceptual level and nociceptive awareness in chronic migraine headache. Conducting a validity and reliability study of the "Fremantle Headache Awareness Questionnaire" developed from The Fremantle Back Awareness Questionnaire in Turkish society can provide objective results in evaluating the effectiveness of treatment as a practical evaluation method in clinics. Hypotheses:

H0: The Fremantle Headache Awareness Questionnaire is not valid and reliable for the Turkish population in chronic migraine patients.

H1: The Fremantle Headache Awareness Questionnaire is valid and reliable for the Turkish population in chronic migraine patients.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with chronic migraine
* Being between the ages of 18-70,
* Being able to read, speak, understand and write Turkish in order to understand the items/questions of the surveys and scales and to give correct answers.

Exclusion Criteria:

* Having any headache diagnosis other than chronic migraine,
* Having a history of any systemic disease such as malignant, inflammatory, acute fracture/infection, surgery, neurological, psychological, rheumatological.
* Having neck or back pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 70 who applied to the Department of Neurology of Mersin University Faculty of Medicine and the Department of Neurology of Gazi University Faculty of Medicine and who were diagnosed with chronic migraine, according to the International Classification of Headache Disorders, 3rd Edition, by a neurologist who is an expert in the field of headache were included in the study.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | In first enrollment, 1 minute
  The visual analog scale consists of the pain level that the person currently experiences with a vertical line on a plane. The pain felt by the person is marked as "0: no pain at all", "10: I feel very severe pain". Scoring is based on the vertical marking the participant makes for the pain he/she marks on the plane with a ruler.
Migraine Disability Assessment Questionnaire | In first enrollment, 3 minutes
  Disability of migraine patients will be assessed with the Migraine Disability Assessment Questionnaire (MEDA). MEDA assesses the last 3 months of disability and consists of a 5-item self-administered test covering disability-related activities at work/school, housework, family, and social or leisure. The total number of days missed in these activities is the total score and classifies disability as minimal disability (0-5 points), mild disability (6-10 points), moderate disability (11-20 points), or severe disability (≥21).
Headache Impact Test-6 | In first enrollment, 3 minutes
  The impact of headache will be assessed with the Headache Impact Test-6 (HIT-6). HIT-6 is a quality of life questionnaire for headaches that assesses vitality, pain, psychological distress, sociability, role, and cognitive functioning. Each item is scored on a 5-point Likert scale (6=never, 8=rarely, 10=sometimes, 11=very often, 13=always). The total score is determined by summing the scores on the six items and ranges from 36 to 78 points. (≤49 = little/no impact, 50-55 = some impact, 56-59 = significant impact, and 60-78 = severe impact; higher scores indicate greater deterioration in quality of life).
Hospital Anxiety and Depression Scale | In first enrollment, 3 minutes
  Anxiety and depression will be assessed with the Hospital Anxiety and Depression Scale (HADS). 7 items of the 14-item scale assess anxiety and 7 items assess depression symptoms. It is scored between 0-3 points. By summing the subscale scores, 0-21 points can be obtained from each of the Depression and Anxiety subscales. It is stated that 0-7 points are the normal range for each subscale, 8-10 points suggest the presence of a mood disorder, and 11 and above points indicate a possible mood disorder. In addition, there are recommended cut-off scores for mild (8-10 points), moderate (11-15) and severe (16 and above) cases.
Pain Catastrophizing Scale | In first enrollment, 3 minutes
  A scale consisting of 13 items that evaluates negative thoughts and feelings about pain experienced. Each item is scored between "0-never and 4-always". The total score of the scale varies between 0-52 and an increase in score indicates a high level of pain catastrophizing. The scale consists of "Helplessness, Magnification, and Rumination" subscales.

CONTACTS AND LOCATIONS:
Locations (13):
- Elite Research and Surgical Hospital, Nicosia, Cyprus
- Turkey (Türkiye) (12):
  - Bozok University, Yozgat, Merkez
  - Gazi University, Ankara, Yenimahalle
  - Mersin University, Mersin, Yenisehir
  - Ankara Atatürk Sanatoryum Training and Research Hospital, Ankara
  - Gazi University, Ankara
  - Gaziantep City Hospital, Gaziantep
  - İstanbul University, Istanbul
  - Silivri State Hospital, Istanbul
  - Kutahya Health Sciences University, Kütahya
  - Headache and Cognition Clinic of Aynur Ozge, Mersin
  - Tokay Gaziosmanpaşa University, Tokat Province
  - Zonguldak Bülent Ecevit University, Zonguldak

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karakas Ugurlu G, Ugurlu M, Erten S, Can SS, Ulusoy Kaymak S, Caykoylu A. Effect of familial Mediterranean fever on sexual and reproductive health in women. Turk J Med Sci. 2017 Apr 18;47(2):463-469. doi: 10.3906/sag-1602-88. PMID 28425232
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Aydemir Ö, Güvenir T, Küey L, Kültür S. Hastane Anksiyete ve Depresyon Ölçeğinin Türkçe formunun geçerlik ve güvenilirlik çalışması. Türk Psikiyatri Dergisi 1997;8(4):280-287
- [Background] Dikmen PY, Bozdag M, Gunes M, Kosak S, Tasdelen B, Uluduz D, Ozge A. Reliability and Validity of Turkish Version of Headache Impact Test (HIT-6) in Patients with Migraine. Noro Psikiyatr Ars. 2020 Apr 24;58(4):300-307. doi: 10.29399/npa.24956. eCollection 2021. PMID 34924791
- [Background] Ertas M, Siva A, Dalkara T, Uzuner N, Dora B, Inan L, Idiman F, Sarica Y, Selcuki D, Sirin H, Oguzhanoglu A, Irkec C, Ozmenoglu M, Ozbenli T, Ozturk M, Saip S, Neyal M, Zarifoglu M; Turkish MIDAS group. Validity and reliability of the Turkish Migraine Disability Assessment (MIDAS) questionnaire. Headache. 2004 Sep;44(8):786-93. doi: 10.1111/j.1526-4610.2004.04146.x. PMID 15330825
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Lai KL, Niddam DM, Fuh JL, Chen WT, Wu JC, Wang SJ. Cortical morphological changes in chronic migraine in a Taiwanese cohort: Surface- and voxel-based analyses. Cephalalgia. 2020 May;40(6):575-585. doi: 10.1177/0333102420920005. Epub 2020 Apr 16. PMID 32299230
- [Background] Onan D, Gokmen D, Ulger O. The Fremantle Neck Awareness Questionnaire in Chronic Neck Pain Patients: Turkish Version, Validity and Reliability Study. Spine (Phila Pa 1976). 2020 Feb 1;45(3):E163-E169. doi: 10.1097/BRS.0000000000003207. PMID 31425430
- [Background] Wand BM, Catley MJ, Rabey MI, O'Sullivan PB, O'Connell NE, Smith AJ. Disrupted Self-Perception in People With Chronic Low Back Pain. Further Evaluation of the Fremantle Back Awareness Questionnaire. J Pain. 2016 Sep;17(9):1001-12. doi: 10.1016/j.jpain.2016.06.003. Epub 2016 Jun 18. PMID 27327235